CLINICAL TRIAL: NCT02300038
Title: Differential Analgesic Effects of Subanesthetic Concentrations of Lidocaine on Spontaneous and Evoked Pain in Human Painful Neuroma
Brief Title: Lidocaine and Neuroma Pain Related Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Adriana Miclescu, MD, PhD, DEAA, Uppsala University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: UppsalaU
Record Dates: First submitted 2014-11-16; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Lidocaine; Sodium Chloride; Salts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Xylocaine) 0.5% (Active Comparator): Injection of 1ml after mixing Lidocaine 10 mg/ml 1 ml +1 ml NaCl was administrated perineuromally
  Interventions: Drug: Lidocaine (Xylocaine); Dietary Supplement: NaCl
- Lidocaine (Xylocaine) 10 mg/ml 0.01% (Placebo Comparator): Injection of 1 ml from 10 mg/ml 1 ml lidocaine Xylocaine +10 ml Nacl was adminsitrated perineuromally
  Interventions: Drug: Lidocaine (Xylocaine); Dietary Supplement: NaCl

INTERVENTIONS:
Drug: Lidocaine (Xylocaine) — perineuromally administration of 1 ml lidocaine
  Other Names: Xylocaine; Lidocaine
Dietary Supplement: NaCl — perineuromally administration of NaCL
  Other Names: Sodium chloride; salt

SUMMARY:
Background Subanesthetics concentrations of lidocaine are able to produce a differential block of the ectopic discharges, but not propagation of impulses, suppressing differentially the associated neuropathic pain symptoms. The aim of this study was to investigate the differences between the analgesic effects of lidocaine 0.5% and a control group of lidocaine 0.1% on several neuroma related pain modalities.

Methods Sixteen patients with neuropathic pain due to painful neuromas caused by nerve injury participated in this randomized, double-blind experiment. The patterns of sensory changes were compared before and after injection of 1 ml lidocaine 0.5% and 0.1% close to the neuroma, the sessions being 1-2 weeks apart. Spontaneous and evoked pains were assessed using a visual analogue scale (VAS), quantitative and qualitative sensory testing.

DETAILED DESCRIPTION:
Patients were recruited by using a postal follow up questionnaire . The number of enrolled subjects in this study- 16 patients, Study design

* The patients visited the Pain Clinic twice.
* The same investigator (AM) performed all study procedure assessments.
* Neuroma was localized by Tinel's sign 14 and when possible (7 patients out of 16), the localization of a neuroma was verified by ultrasound.

Administration of study drug The patients were randomized by a computer generated random list to receive either 1ml lidocaine 0.5% (A) or 1 ml 0.1% (B-control) injected perineuromally.

Pain assessments Duration of the present pain condition was recorded. The patients were asked to rate the mean, maximum, minimum pain intensity of their spontaneous and evoked pain in the week prior to both visits. The pain score was measured from baseline until 60 min after injection. Assessments of pain were done post injection at 15 s, 30 s, 1 min, and at 5-min intervals for the first 30-min post injection and then every 10-min to 1 hr post injection. The assessments of pain were performed between the limbs in the following order: spontaneous pain, then assessment of dynamic mechanical allodynia and then pinprick hyperalgesia.

Spontaneous pain Evaluation of sensory function was performed in the affected limb using bedside examination according to EFNS (European Federation of Neurological Societies)guidelines: light touch, pinprick sense, warmth (40°) and cold (25°) temperature stimuli were tested.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* with a history of persistent spontaneous and/or evoked pain (by e.g. touch, movement),
* who scored an average daily pain intensity of at least 4 on a 0-10 point numerical pain scale (NRS) interfering with daily activities and who had pain at least 3 months duration.
* They all had neuromas after upper extremity surgery or other trauma affecting the radial, ulnar, median or digital nerves and were eligible to participate in the study after giving written informed consent.

Exclusion Criteria:

* Patients with other conditions that might confound assessment of pain attributed to posttraumatic upper limb pain or
* any condition/disease that could interfere with the study measurements, such as drug abuse, diabetes, vascular disease, polyneuropathy or psychiatric diseases were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2013-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The primary end-point measure was defined as the change in pain score measured from baseline until 60 min after injection | 60 min